CLINICAL TRIAL: NCT06391580
Title: A Multi-center, Randomized, No-treatment Controlled, Evaluator-blinded, Superiority Clinical Trial to Evaluate the Efficacy and Safety of LANLUMA V to Improve Jawline Contour Deficit
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of LANLUMA V to Improve Jawline Contour Deficit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinclair Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDM6010A-301
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Jawline Contour Deficit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poly-L-lactin Acid (PLLA) Based Facial Injectable (Experimental): Poly-L-lactin Acid (PLLA) Based Facial Injectable
  Interventions: Device: Poly-L-lactin Acid (PLLA) Based Facial Injectable
- No treatment control (No Intervention): No treatment control

INTERVENTIONS:
Device: Poly-L-lactin Acid (PLLA) Based Facial Injectable — Poly-L-lactin Acid (PLLA) Based Facial Injectable
  Arms: Poly-L-lactin Acid (PLLA) Based Facial Injectable

SUMMARY:
A Multi-center, Randomized, No-treatment Controlled, Evaluator-blinded, Superiority Clinical Trial to Evaluate the Efficacy and Safety of LANLUMA V to Improve Jawline Contour Deficit

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who aged 18 years or older (subject to the date of signing the informed consent), male or female;
2. Subjects with a MJAS score of moderate to severe levels (2~3 scores) in terms of bilateral jawline contour as evaluated by the blinded evaluator, and the scores of bilateral jawline contour must meet the criteria but not required to be the same;
3. Subjects who are seeking to receive corrective treatment for jawline contouring;
4. Subjects who are in good health and suitable to receive corrective treatment for jawline contouring as evaluated by the blinded evaluator;
5. Subjects who voluntarily sign the ICF, understand and accept the study duration, and are able to comply with all requirements including treatment, follow-ups and other study procedures as scheduled;

Exclusion Criteria:

1. Subjects with non-aging skin laxity and lipoatrophy which may affect the evaluation of efficacy in the midface or mandibular region as identified by the investigator;
2. Subjects who are known to be allergic to any local anesthetics (such as lidocaine or other amide anesthetics), or have a history of severe allergic reactions or anaphylactic shock;
3. Subjects who have residual defects, scars, deformities, tattoos, perforations, hair, unhealed wounds, active skin diseases or inflammations (such as eczema, acnes, psoriasis, and herpes zoster), abscesses, carcinogenesis or precancerous lesions and other conditions that may affect evaluation of vision and efficacy or increase the risk of treatment in the injection and evaluation areas;
4. Subjects with unstable and/or irreproducible malocclusion, or bruxism, hypertrophy or asymmetry of masseter, lockjaw, active temporomandibular disorders or active periodontal diseases;
5. Subjects who have a tendency to develop keloids, hypertrophic scars, or any other healing disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy rate of jawline contour deficit improvement in the test group at 48 weeks after the last injection and that in the control group at 48 weeks after randomization, evaluated by blinded evaluators using the MJAS. | 48 weeks

SECONDARY OUTCOMES:
Efficacy rate of jawline contour deficit improvement (as evaluated by blinded evaluators, except for the primary efficacy index visit point) | 5, 12, 24 and 36 weeks
Jawline contour deficit improvement score (as evaluated by blinded evaluators) | 5, 12, 24, 36 and 48 weeks
Change in FACE-QTM Satisfaction with Lower Face and Jawline score from the baseline (as evaluated by the subject) | 5, 12, 24 36 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hongyi Zhao, Principal Investigator — Beijing Hospital, China
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No